CLINICAL TRIAL: NCT04492618
Title: Ruxolitinib Cream in the Treatment of Cutaneous Necrobiosis Lipoidica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron R. Mangold (Other)
Responsible Party: Sponsor-Investigator, Aaron R. Mangold, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-004087
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Necrobiosis Lipoidica
MeSH Terms: conditions — Necrobiosis Lipoidica | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Necrobiosis Lipoidica (Experimental): Adults with cutaneous Necrobiosis Lipoidica (NL) up to 10% of the body surface area (BSA) treated with Ruxolitinib cream
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib cream 1.5%, topical application will be used twice daily on lesions of Necrobiosis Lipoidica

SUMMARY:
This research study is evaluating the safety and efficacy of a topical drug treatment "Ruxolitinib" in treating Necrobiosis Lipoidica (NL).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and comply with the requirements of the study and communicate with the investigator. Subjects must give written, signed, and dated informed consent before any study related activity is performed. When appropriate, a legal representative will sign the informed consent according to local laws and regulation
* Both men and women must be at least 18 years of age at the time of screening
* Subjects must have clinical and histological features of NL
* Subjects must have at least one NL lesion measuring at least 1.7 cm
* NL must not affect greater than 10% BSA

Exclusion Criteria:

* On excluded therapies, not on a stable dose of a therapy, or incompletely washed out for a therapy (Table-1).
* Known hypersensitivity to Ruxolitinib formulation.
* Pregnant or nursing (lactating) women (pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test).
* Women of childbearing potential [Post-menopausal or not of child-bearing potential is defined by: 1 year of natural (spontaneous) amenorrhea or Surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks ago. Oophorectomy alone must be confirmed by follow up hormone level assessment to be considered not of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using medically acceptable methods of contraception which includes:

  * Total abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception).
  * Female sterilization (bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. Oophorectomy alone requires follow up hormone level assessment for fertility.
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
  * Barrier methods of contraception: condom or occlusive cap.
  * Use of oral, injected or implanted hormonal methods of contraception or other forms or hormonal contraception that have complete efficacy (failure <1%). (The dose of the contraceptive should be stable for 3 months).
* Active ongoing inflammatory diseases of the skin other than NL that might confound the evaluation of the benefit of ruxolitinib cream.
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions) which, in the opinion of the investigator, significantly immunocompromised the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
* Active systemic infections during the 2 weeks prior to randomization (common cold viruses not included) or any infection that reoccurs on a regular basis.
* Current severe progressive or uncontrolled disease which the investigator renders the subject unsuitable for the trial or puts the subject at increased risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Mangold, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Necrobiosis Lipoidica: Adults with cutaneous Necrobiosis Lipoidica (NL) up to 10% of the body surface area (BSA) were treated with Ruxolitinib cream
  Ruxolitinib: Ruxolitinib cream 1.5%, topical application was used twice daily on lesions of Necrobiosis Lipoidica
Period: Overall Study
Arm/Group | Necrobiosis Lipoidica
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Necrobiosis Lipoidica
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Necrobiosis Lipoidica (NL) Lesion Score
Description: The NL skin scoring system examines the index treatment lesion on a scale from 0 (none) to 3 (severe) for each of the following areas: erythema, infiltration, ulceration, and pain. A total possible score of 0-12, with lower scores indicating none and higher scores indicating more severe.
Time Frame: Baseline, week 12
Population: 1 Subject withdrew. Week 12 data was not collected nor analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Necrobiosis Lipoidica
Number analyzed (Participants) | 11
score on a scale | -2.7 (1.6)
Statistical Analysis 1: Comparison: Necrobiosis Lipoidica; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all subjects from baseline to end of study, approximately 16 weeks.
Arm/Group | Necrobiosis Lipoidica
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Necrobiosis Lipoidica (N=12)
Abdominal pain (Gastrointestinal disorders) | 1
Basal cell carcimona removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Burning sensation (Skin and subcutaneous tissue disorders) | 1
Burning sensation on NL spots (Skin and subcutaneous tissue disorders) | 1
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Heaviness Bilateral legs (Musculoskeletal and connective tissue disorders) | 1
Heightened sensitivity on lesions (Skin and subcutaneous tissue disorders) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Lower extremity aches (Musculoskeletal and connective tissue disorders) | 1
Nausea (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Tingling feeling left shin (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT04492618/Prot_SAP_000.pdf